CLINICAL TRIAL: NCT02740959
Title: Effects of PG2 on Fatigue-Related Symptom Clusters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Chia-Chin Lin, Dean, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N201509006
Record Dates: First submitted 2016-02-16; First posted 2016-04-15 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Cancer-related Fatigue
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astragalus Polysaccharides 500 mg (Experimental): PG2 (500 mg in 500 ml saline), t.i.w. via i.v. infusion for 2.5-3.5 hours over 2 treatment cycles (8 weeks)
  Interventions: Drug: Astragalus Polysaccharides 500 mg
- Astragalus Polysaccharides 250 mg (Experimental): PG2 (250 mg in 500 ml saline), t.i.w. via i.v. infusion for 2.5-3.5 hours over 2 treatment cycles (8 weeks)
  Interventions: Drug: Astragalus Polysaccharides 250 mg

INTERVENTIONS:
Drug: Astragalus Polysaccharides 500 mg — PG2 Injection 500 mg PG2 (500 mg in 500 ml saline), t.i.w. via i.v. infusion for 2.5-3.5 hours over 2 treatment cycles (8 weeks)
  Other Names: PG2 Injection 500 mg PG2 (500 mg in 500 ml saline)
  Arms: Astragalus Polysaccharides 500 mg
Drug: Astragalus Polysaccharides 250 mg — PG2 Injection 250 mg PG2 (250 mg in 500 ml saline), t.i.w. via i.v. infusion for 2.5-3.5 hours over 2 treatment cycles (8 weeks)
  Other Names: PG2 Injection 250 mg PG2 (250 mg in 500 ml saline)
  Arms: Astragalus Polysaccharides 250 mg

SUMMARY:
This study is for an "add-on" study to the "main" study (Protocol No.: PH-CP012). The information of patients from main study will be collected by questionnaire survey and actigraphy measurement to evaluate the relationship between fatigue, depression and sleep disorder and the efficacy of PG2 after treatment.The association between symptom cluster and circadian rhythm will be also further explored.

DETAILED DESCRIPTION:
The study is "PG2 Treatment for Improving Fatigue among Advanced Cancer Patients under Standard Palliative Care" (Protocol Number: PH-CP012) of the additional plan, through questionnaires and using actigraphy measuring circadian rhythm collect patient data master plans, assessed for "PG2" treatment of cancer patients before and after treatment fatigue, depression, sleep disorders and other related symptoms of resistance and the effectiveness of treatment, and to further explore the symptom clusters in cancer patients associated with the circadian rhythm

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the informed consent form
* The age of eligible patients should be 20 years old.
* Eligible patients must have locally advanced or metastatic cancer or inoperable advanced cancer.
* Patients are under standard palliative care (SPC) at hospice setting and have no further curative options available.
* Patients with BFI fatigue score 4 during screening.
* Patients have a life expectancy of at least 3 months as determined by the investigator.
* Patient must be willing and able to complete quality of life questionnaires.

Exclusion Criteria:

* Female patients are pregnant or breast-feeding.
* Patients with uncontrolled systemic disease such as active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus.
* Patients take central nervous system stimulators such as Methylphenidate within 30 days before screening.
* Patients have enrolled or have not yet completed other investigational drug trials within 30 days before screening.
* Patients with Karnofsky Performance Scores less than 30 % at time of screening
* Patients who are diagnosed as dying status

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Scale | about 5-10 minutes
Hospital Anxiety and Depression Scale | about 5-10 minutes
Actigraphy measuring circadian rhythm | 3-month course of treatment, a total of three measurements, each measurement 7 days
  three measurements means:3 days prior to the first dose of study medication began wearing courses of the last visits to the first week; last treatment of 3rd and 7th weeks of medication visits began wearing last time between the 4th and 8th week of visits

CONTACTS AND LOCATIONS:
Overall Officials: Lin C Chin, PhD., RN, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University -Shung Ho Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No